CLINICAL TRIAL: NCT06313866
Title: the Clinical Effect of TCM Sniffing Therapy Combined With Electroacupuncture in the Treatment of Cognitive Impairment After Stroke
Brief Title: the Clinical Effect of TCM Sniffing Therapy Combined With Electroacupuncture in PSCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024ZL368
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Smell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- control (No Intervention): Donepezil hydrochloride was administered at 5 mg once a day (nightly) for 30 days without adverse reactions and then increased to 10 mg once a day (nightly) for 4 weeks.
- Electronuchal acupuncture group treatment (Experimental): Use the neck needle to take the Fengchi and Gongxue on both sides (1.5cm directly below Fengchi point).
  Interventions: Dietary Supplement: control; Other: Electronuchal acupuncture group treatment
- Smell therapy group treatment (Experimental): The volatile oil of Acorus calamus is packed in the sniffer. Smell at the sniffing end, breathe evenly, 5-10 minutes each time, 3-5 times a day, for a total of 4 weeks of treatment.
  Interventions: Dietary Supplement: control; Other: Smell therapy group treatment
- The combined treatment (Experimental): The electro-neuchal acupuncture combined with sniffing and suction therapy group is treated with sniffing and suction therapy on the basis of electro-neuchal acupuncture treatment.
  Interventions: Dietary Supplement: control; Other: Electronuchal acupuncture combined with smell and inhalation therapy group treatment
- normal (Other): The volatile oil of Acorus calamus is packed in the sniffer. Smell at the sniffing end, breathe evenly, 5-10 minutes each time, 3-5 times a day, for a total of 4 weeks of treatment.
  Interventions: Other: Smell therapy group treatment
- Sham group (Sham Comparator): In the sham stimulation group, non-transdermal comfortable acupuncture will be used to make the patients experience a feeling similar to acupuncture.
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Dietary Supplement: control — Donepezil hydrochloride was administered at 5 mg once a day (nightly) for 30 days without adverse reactions and then increased to 10 mg once a day (nightly) for 4 weeks.
  Arms: Electronuchal acupuncture group treatment; Smell therapy group treatment; The combined treatment
Other: Electronuchal acupuncture group treatment — Electronuchal acupuncture
  Arms: Electronuchal acupuncture group treatment
Other: Smell therapy group treatment — nasal suction intervention with volatile oil of Acorus calamus
  Arms: Smell therapy group treatment; normal
Other: Electronuchal acupuncture combined with smell and inhalation therapy group treatment — On the basis of electric nuchal acupuncture treatment, sniffing and inhalation therapy is given.
  Arms: The combined treatment
Other: Sham stimulation — In the sham stimulation group, non-transdermal comfortable acupuncture will be used to make the patients experience a feeling similar to acupuncture.
  Arms: Sham group

SUMMARY:
The patients with cognitive impairment after stroke were divided into control group, electroacupuncture group, olfactory therapy group, electroacupuncture combined with olfactory therapy group, and sham group with 35 people in each group. After the end of the treatment, the clinical efficacy was evaluated.

DETAILED DESCRIPTION:
The patients with cognitive impairment after stroke were divided into control group, electroacupuncture group, olfactory therapy group, and electroacupuncture combined with olfactory therapy group, and sham group with 35 people in each group. All patients were treated with conventional drugs and general supportive treatment, and on the basis of this, the electroacupuncture group was given electroacupuncture treatment at bilateral Fengchi and Gongxue, the smell suction therapy group was given the intervention of volatile oil nasal suction of Acorus calamus, and the electroacupuncture group combined with smell and suction therapy group was given electroacupuncture treatment at the same time as the electroacupuncture treatment of bilateral Fengchi and Gongxue. In the sham stimulation group, non-transdermal comfortable acupuncture will be used to make the patients experience a feeling similar to acupuncture. After the 1 month innervation,the main efficacy indicators: Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Barthel Index (MBI) score, and the secondary efficacy indicators: Transcranial Doppler (TCD), near-infrared functional brain imaging , magnetic resonance examination， the heart rate,blood pressure and the State Trait Anxiety Inventory （STAI）are collected.

ELIGIBILITY:
Inclusion Criteria:

* (1) Stroke as per the TCM definition, presenting symptoms include unilateral paresis or paralysis, sensory deficits, speech impairment, and hemianopsia. PSCI diagnosis involves clinically significant deficits in at least one cognitive domain and severe disruption of instrumental ADLs/ADLs.; (2) The scores on the MMSE scale must adhere to the following criteria: Less than 17 points for individuals with illiteracy, less than 20 points for those with primary school education, and less than 24 points for individuals with a middle school education or higher.; (3) Aged under 70 years; (4) No history of mental illness, clear consciousness, stable vital signs, and able to complete the scale assessment; (5) Within 6 months post-stroke, diagnosed as a patient in the recovery period of cerebral infarction (or cerebral hemorrhage) at admission; (6) Signed informed consent by the patient or their family.

Exclusion Criteria:

* (1) Transient ischemic attack; (2) Subarachnoid hemorrhage; (3) History of severe liver or kidney diseases, mental illness, epilepsy, asthma, or obstructive pulmonary diseases; (4) Occurrence of cognitive impairment prior to stroke; (5) Severe communication barriers; (6) Substance abuse or heavy alcohol consumption; (7) Implanted cardiac pacemakers or other electronic devices.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
MoCA | 0,4 weeks after the intervention, 8 weeks after the intervention
  Montreal Cognitive Assessment Scale

SECONDARY OUTCOMES:
MMSE | 0,4 weeks after the intervention,8 weeks after the intervention
  Mini-Mental State Examination
MBI | 0,4 weeks after the intervention,8 weeks after the intervention
  Barthel index score
TCD | 0,4 weeks after the intervention
  Transcranial Doppler examination
Near-infrared functional imaging of the brain | 0,4 weeks after the intervention
  Near-infrared functional imaging of the brain
Magnetic resonance scanning | 0,4 weeks after the intervention
  Magnetic resonance scanning
the State Trait Anxiety Inventory (STAI) | 0,4 weeks after the intervention
  the State Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Xinyun Li, doctor, Principal Investigator — hangzhou medical colleage
Locations (1):
- the Affiliated Zhejiang Provincial People's Hospital to Hangzhou Medical College., Hangzhou, Zhejiang, China